CLINICAL TRIAL: NCT02639793
Title: A Nationwide Multicenter Trial Assessing the Effects of Catheter Ablation on Burden of Atrial Fibrillation Recorded by Implantable Cardiac Monitor
Brief Title: Effects of Catheter Ablation on Burden of Atrial Fibrillation (MRICEMAN)
Acronym: MRICEMAN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heikki Huikuri (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Sponsor-Investigator, Heikki Huikuri, Professor, University of Oulu
Organization: University of Oulu (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFOulu
Record Dates: First submitted 2015-12-09; First posted 2015-12-24 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Atrial Fibrillation
Keywords: arrhythmias, quality of life
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- manual radiofrequency ablation (Active Comparator): Radiofrequency catheter ablation using manual catheter manipulation will be used as an ablation technique.
  Interventions: Procedure: catheter ablation
- magnet navigation ablation (Active Comparator): Radiofrequency catheter ablation using remote magnet navigation will be used as an ablation technique.
  Interventions: Procedure: catheter ablation
- cryoablation (Active Comparator): Catheter ablation using cryoablation technique will be used as an ablation technique of atrial fibrillation.
  Interventions: Procedure: catheter ablation

INTERVENTIONS:
Procedure: catheter ablation — Three different catheter ablation techniques will be used aimed at isolating the pulmonary veins from left atrium.The endpoint is defined as absence or dissociation of all pulmonary vein potentials as confirmed by the circular mapping catheter after a waiting period of 30 minutes after the last ablation. The use of adenosine or isoproterenol to detect concealed pulmonary vein conduction is voluntary.

SUMMARY:
The study will assess the atrial fibrillation burden recorded By implantable loop recorder at 12 and 24 months compared to baseline. The patients with clinical indication fo catheter ablation of paroxysmal atrial fibrillation will be randomized to three techniques: manual radiofrequency ablation, radiofrequency ablation using remote magnet monitoring, and cryoablation.

DETAILED DESCRIPTION:
A total of 300 patients will be randomized to three different catheter ablation techniques (100 patients/group); radiofrequency ablation using remote magnet navigation, radiofrequency ablation using manual method, and cryoablation. A loop recorder (REVEAL) is implanted one month before the catheter ablation of paroxysmal atrial fibrillation and the effects of atrial fibrillation burden will be compared between the three methods at 12 and 24 months after ablation excluding the first three months´ blanking period.

The primary endpoints are:

1. the proportion of patients remaining free from atrial fibrillation, atrial flutter or atrial tachycardia (> 2 minutes) recorded by the implantable cardiac monitor (Medtronic) at 24 months follow-up and
2. total atrial fibrillation burden recorded by the loop recorder.

Other endpoints:

1. Atrial fibrillation burden in 7 days Holter recording at 12 and 24 months compared to baseline,
2. the time to first documented symptomatic and asymptomatic recurrence of atrial fibrillation
3. prescription of antiarrhythmic drugs after the 3 months blanking period following the ablation
4. re-ablation after the index ablation procedure,
5. total procedural duration;
6. total time of fluoroscopy and radiation dose;
7. number and duration of cardiovascular hospitalization;
8. quality of life questionnaires at 12 months and 24 month compared with baseline,
9. cognitive function at 12 and 24 month compared with baseline,
10. cost-efficacy of the different ablation techniques.

ELIGIBILITY:
Inclusion criteria:

* Patients with symptomatic paroxysmal atrial fibrillation fulfilling the contemporary guideline criteria for AF ablation

Exclusion Criteria:

- Any contraindication to catheter ablation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Free of atrial fibrillation | 24 months
  the proportion of patients remaining free from AF, atrial flutter (AFL) or atrial tachycardia (AT) (> 2 minutes) recorded by the implantable cardiac monitor (ICM, Reveal, Medtronic Co.) at 24 months.

SECONDARY OUTCOMES:
Total AF burden | 24 months
  total AF burden recorded by the implantable loop recorder during the 24 month follow-up.
Incidence of adverse events | 24 months
  Safety is one of the secondary endpoints. The following potential adverse events will be monitored: Any previous left atrial ablation or surgery Any cardiac surgery or percutaneous coronary intervention within three months prior to enrolment.
  Secondary AF Stroke or transient ischemic attack within six months prior to enrolment Myocardial infarction within three months prior to enrolment Left ventricular ejection fraction < 40 % Anteroposterior left atrial diameter >55 mm by transthoracic or transesophageal echocardiography Implanted prosthetic valve

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Huikuri, Prof, Principal Investigator — University of Oulu
Locations (2):
- Finland (2):
  - UOulu, Oulu
  - Heikki Huikuri, Oulu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: wep-page — http://www.oulu.fi/yliopisto